CLINICAL TRIAL: NCT05065827
Title: Lung Ultrasound Findings in Patients With COVID-19 in a UK Emergency Department
Brief Title: Lung Ultrasound Findings in Patients With COVID-19 in a UK ED
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C&W20/050; IRAS number 286642 (Other: Integrated Research Application System)
Record Dates: First submitted 2021-09-30; First posted 2021-10-04 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Coronavirus; Corona Virus Infection; SARS-CoV Infection
Keywords: COVID-19; Lung ultrasound; Retrospective
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal oxygenation: Normal oxygenation based on the BERLIN criteria for ARDS
- Mild deficit in oxygenation: Mild deficit in oxygenation based on the BERLIN criteria for ARDS
- Moderate deficit in oxygenation: Moderate deficit in oxygenation based on the BERLIN criteria for ARDS
- Severe deficit in oxygenation: Severe deficit in oxygenation based on the BERLIN criteria for ARDS

SUMMARY:
The investigators aim to carry out a retrospective observational study, analysing lung ultrasound images from patients who have presented to A&E for routine diagnostic purposes (ruling out cardiogenic pulmonary oedema, Pulmonary embolism and pericardial effusions) and systematically assessing for abnormalities typical for COVID-19 infection (Pleural irregularities, B lines, consolidations, pleural effusions). Doing this, the investigators will also develop a suggestion for a standardised technique for lung ultrasound which can be transferred to other clinical settings (Intensive Care, Acute medical Unit) and could form the basis for an international standard. Thirdly, the investigators aim to correlate our findings to clinical severity judged by oxygenation status on arrival in ED. To the investigators' knowledge, this is the first study of this kind.

DETAILED DESCRIPTION:
COVID-19 is a new disease significant morbidity and mortality which has reached pandemic status. Due to its highly contagious nature, is essential to characterise the disease pathology quickly and reliably. The lung changes that can be seen in patients with COVID-19 can precede clinical symptoms and are picked up on ultrasound more reliably than on conventional chest XR. In addition, ultrasound is devoid of harmful radiation, is quick to perform, and easily learned by doctors who routinely use ultrasound such as in the Emergency Department. To date, there is no data systematically analysing the ultrasound changes in COVID-19 and relating this to disease severity. The data from our study will be contribute significantly to developing strategies for safe triage with regards to cohorting, diagnosis and prognosis of COVID-19.

In this research study, lung ultrasound scans will be retrospectively analysed that were obtained from patients who presented to the emergency department during March-May 2020 with shortness of breath, who were subsequently diagnosed with COVID-19 either by PCR test or composite diagnostic criteria of lymphopenia and positive Chest XR or CT scan report.

The lung ultrasound images will be retrospectively scored for the presence of absence of 5 lung abnormalities (pleural irregularity, B lines, small peripheral consolidation, large consolidation, small effusion (<1cm) and large effusion (>1cm). Scoring will be performed by 2 independent observers with experience in lung ultrasound. In addition, each abnormality will be analysed for preferential location within the lung.

The patients will be grouped into 4 groups of clinical severity (normal oxygenation, mild, moderate and severe deficit in oxygenation) based on the BERLIN criteria for ARDS, and lung abnormalities as seen on lung ultrasound will be analysed for correlation to clinical severity.

ELIGIBILITY:
Inclusion Criteria:

* Presented to the ED between March-May 2020 with dyspnoea
* COVID-19 positive either by PCR test or composite diagnostic criteria of lymphopenia and positive Chest XR report
* Received lung ultrasound as part of investigations during ED attendance

Exclusion Criteria:

* < 18 years of age
* Not diagnosed with COVID-19

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with COVID-19 viral infection.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Characterisation of lung changes in COVID-19 patients as seen on ultrasound | 2-3 months
  Retrospective scoring of lung ultrasound images (12-zone ultrasound where clinical status allowed) for each of 5 lung abnormalities (pleural irregularity, B lines, small peripheral consolidation, large consolidation, small effusion (<1cm) and large effusion (>1cm).
  The images will be scored by 2 independent observers and the scores will be analysed based on the occurrence, location within the lung and clinical correlation

SECONDARY OUTCOMES:
Correlation of lung changes as seen on ultrasound with clinical severity as per the Berlin ARDS criteria | 2-3 months
  Patients will be grouped into 4 groups of clinical severity (normal oxygenation, mild, moderate and severe deficit in oxygenation) based on the BERLIN criteria for ARDS.
  The data will be analysed by standard statistical tests comparing binomial data between unpaired and paired groups, as well as comparing more than three unmatched groups. This will include Chi-square, McNemar and paired t-tests and one-way ANOVA tests

CONTACTS AND LOCATIONS:
Overall Officials: Paramjeet Deol, MBChB FRCEM, Principal Investigator — paramjeet.deol@chelwest.nhs.uk
Locations (1):
- Chelsea and Westminster Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A, Barre O. The comet-tail artifact. An ultrasound sign of alveolar-interstitial syndrome. Am J Respir Crit Care Med. 1997 Nov;156(5):1640-6. doi: 10.1164/ajrccm.156.5.96-07096. PMID 9372688
- [Background] Lichtenstein D. Lung ultrasound in the critically ill. Curr Opin Crit Care. 2014 Jun;20(3):315-22. doi: 10.1097/MCC.0000000000000096. PMID 24758984
- [Background] Lichtenstein DA. Current Misconceptions in Lung Ultrasound: A Short Guide for Experts. Chest. 2019 Jul;156(1):21-25. doi: 10.1016/j.chest.2019.02.332. Epub 2019 Mar 11. No abstract available. PMID 30872018
- [Background] Soldati G, Smargiassi A, Inchingolo R, Buonsenso D, Perrone T, Briganti DF, Perlini S, Torri E, Mariani A, Mossolani EE, Tursi F, Mento F, Demi L. On Lung Ultrasound Patterns Specificity in the Management of COVID-19 Patients. J Ultrasound Med. 2020 Nov;39(11):2283-2284. doi: 10.1002/jum.15326. Epub 2020 May 8. No abstract available. PMID 32383781
- [Background] Vetrugno L, Bove T, Orso D, Barbariol F, Bassi F, Boero E, Ferrari G, Kong R. Our Italian experience using lung ultrasound for identification, grading and serial follow-up of severity of lung involvement for management of patients with COVID-19. Echocardiography. 2020 Apr;37(4):625-627. doi: 10.1111/echo.14664. Epub 2020 Apr 15. PMID 32239532
- [Background] Volpicelli G, Gargani L. Sonographic signs and patterns of COVID-19 pneumonia. Ultrasound J. 2020 Apr 21;12(1):22. doi: 10.1186/s13089-020-00171-w. PMID 32318891
- [Background] Xing C, Li Q, Du H, Kang W, Lian J, Yuan L. Lung ultrasound findings in patients with COVID-19 pneumonia. Crit Care. 2020 Apr 28;24(1):174. doi: 10.1186/s13054-020-02876-9. No abstract available. PMID 32345353
- [Background] Yasukawa K, Minami T. Point-of-Care Lung Ultrasound Findings in Patients with COVID-19 Pneumonia. Am J Trop Med Hyg. 2020 Jun;102(6):1198-1202. doi: 10.4269/ajtmh.20-0280. PMID 32333544
- [Background] Soldati G, Smargiassi A, Inchingolo R, Buonsenso D, Perrone T, Briganti DF, Perlini S, Torri E, Mariani A, Mossolani EE, Tursi F, Mento F, Demi L. Proposal for International Standardization of the Use of Lung Ultrasound for Patients With COVID-19: A Simple, Quantitative, Reproducible Method. J Ultrasound Med. 2020 Jul;39(7):1413-1419. doi: 10.1002/jum.15285. Epub 2020 Apr 13. PMID 32227492
- [Background] Ferguson ND, Fan E, Camporota L, Antonelli M, Anzueto A, Beale R, Brochard L, Brower R, Esteban A, Gattinoni L, Rhodes A, Slutsky AS, Vincent JL, Rubenfeld GD, Thompson BT, Ranieri VM. The Berlin definition of ARDS: an expanded rationale, justification, and supplementary material. Intensive Care Med. 2012 Oct;38(10):1573-82. doi: 10.1007/s00134-012-2682-1. Epub 2012 Aug 25. PMID 22926653